CLINICAL TRIAL: NCT02994979
Title: Multicomponent Intervention to Prevent Delirium in Nursing Homes
Brief Title: Nursing Assistant Intervention to Prevent Delirium in Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jewish Home & Hospital Lifecare System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2016-04
Record Dates: First submitted 2016-12-09; First posted 2016-12-16 (Estimated); Results first posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Delirium-prevention group (Experimental): Multicomponent delirium prevention intervention led by a Certified Nursing Assistant (CNA) adapted for the long-term care setting from the Hospital Elder Life Program.
  Interventions: Other: Delirium-prevention
- Usual care group (Sham Comparator): Usual care plus a sham visit from the intervention CNA
  Interventions: Other: Sham comparator

INTERVENTIONS:
Other: Delirium-prevention — Patients will be seen by an intervention CNA at least once daily 7 days a week. The CNA will be English/Spanish bilingual and will provide intervention components guided by structured protocols and a daily visit form. A typical visit lasts 30 minutes and begins with an introduction and orientation activity followed by provision of water, a reminiscence activity or game, a physical exercise, and a snack and second cup of water. Patients may also receive a relaxation visit at night and given a warm drink, a hand or foot massage, and quiet music. Daily visits will last for the duration of the illness and 7 days following the illness end. Illness end is defined as the last day of illness treatment (e.g., last day of antibiotics) or monitoring (e.g., last day on nursing "24-hour report"). During weekly intervention staff meetings patients will be discussed with the primary medical and nursing team. The planned intervention group sample size results in a case load of 4-8 patients.
  Other Names: HELP-LTC
  Arms: Delirium-prevention group
Other: Sham comparator — Usual care plus sham visits by CNA
  Arms: Usual care group

SUMMARY:
Delirium is an acute confusion that occurs in one third of hospitalized older adults. As compared to those without delirium, hospitalized patients with delirium have longer hospital stays, higher mortality, and increased risk of nursing home utilization. Substantial attention has been paid to developing, testing, and disseminating interventions to prevent delirium in the hospital but, to date, not in the nursing home setting. In a previous study we used known information on delirium risk factors to develop an intervention that can be delivered at onset of acute illness in nursing home patients. The current study is designed to test the effect of this intervention in a single-site clinical trial. Objectives: 1) to determine, as compared to control, the effect of a multicomponent intervention targeting delirium risk factors on delirium frequency, delirium severity, cognitive and physical function decline, and hospitalization in nursing home patients with acute illness, and 2) to identify features of the intervention associated with occurrence of delirium and other outcomes. Approach: We will screen nursing home patients on 17 long-term care units at a large, urban nursing home who experience onset of a change in condition according to established criteria, and enroll and assign them to intervention or control in a 1:1 ratio. Those assigned to intervention will receive daily visits from an Elder Life Specialist, a mobile Certified Nursing Assistant trained to provide services to counter risks for delirium, including dehydration, immobility, cognitive impairment, undernutrition, and sleep problems, for the duration of the acute illness and for 1 week following. Patients assigned to control will receive usual care from the unit-based nurses and the patient's primary team. Delirium will be assessed 5 days a week by a research assistant. Cognitive and physical function decline and hospital transfer will be ascertained during a 1 month follow-up period. We will compare outcomes between intervention and control, as well as examine associations between outcomes and intervention features such as number and duration of visits.

DETAILED DESCRIPTION:
Delirium is an acute cognitive disorder with features of inattention, disorganized thinking, and disordered consciousness that occurs in one third of hospitalized older adults. As compared to those without delirium, hospitalized patients with delirium have longer hospital stays, higher mortality, and increased risk of nursing home utilization. Substantial attention has been paid to developing, testing, and disseminating interventions to prevent delirium in the hospital but, to date, not in the nursing home setting. In a previous study we used known information on delirium risk factors to develop a multicomponent intervention that can be delivered at onset of acute illness in nursing home patients. We demonstrated the intervention's feasibility, adherence, and acceptance by patients and staff. The current study is designed to test the efficacy of this intervention in a single-site cluster-randomized trial. Objectives: 1) to determine, as compared to control, the effect of a multicomponent intervention targeting delirium risk factors (immobility, cognitive impairment, dehydration, undernutrition, sleep, and medication use) on the primary outcome of delirium frequency in nursing home patients with acute illness, and the secondary outcomes of delirium severity, cognitive and physical function decline, and hospitalization associated with acute illness, and 2) to identify features of the intervention, including "dose" and components, associated with occurrence of delirium and its severity, cognitive and physical function decline, and hospitalization associated with acute illness. Approach: We will screen nursing home patients on 17 long-term care units at a large, urban nursing home who experience onset of an acute change in condition according to established criteria, and enroll and assign them to intervention or control in a 1:1 ratio. Those assigned to intervention will receive daily visits from an Elder Life Specialist, a mobile Certified Nursing Assistant trained to provide services to counter risks for delirium, including dehydration, immobility, cognitive impairment, undernutrition, and sleep problems, for the duration of the acute illness and for 1 week following, in collaboration with the patient's primary medical and nursing team. Patients assigned to control will receive usual care from the unit-based nurses and the patient's primary team. Delirium will be assessed 5 days a week by a research assistant blinded to study hypotheses and group assignment. Cognitive and physical function decline and hospital transfer will be ascertained during a 1 month follow-up period. We will conduct analyses to compare outcomes between intervention and control, as well as examine associations between outcomes and intervention features such as number and duration of visits.

ELIGIBILITY:
Inclusion Criteria

* Long-term care nursing home resident at The New Jewish Home
* Acute change in condition or just returned from the hospital
* Assent to participate in study

Exclusion Criteria

* Discharge or death expected before 2 months
* Nonverbal or unable to follow simple commands

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2016-11; Primary Completion 2018-08-21 (Actual); Study Completion 2018-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Boockvar, MD, Principal Investigator — Mount Sinai School of Medicine; The New Jewish Home
Locations (1):
- The New Jewish Home, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Delirium-prevention Group: Multicomponent delirium prevention intervention led by a Certified Nursing Assistant (CNA) adapted for the long-term care setting from the Hospital Elder Life Program.
  Delirium-prevention: Patients will be seen by an intervention CNA at least once daily 7 days a week. The CNA will be English/Spanish bilingual and will provide intervention components guided by structured protocols and a daily visit form. A typical visit lasts 30 minutes and begins with an introduction and orientation activity followed by provision of water, a reminiscence activity or game, a physical exercise, and a snack and second cup of water. Patients may also receive a relaxation visit at night and given a warm drink, a hand or foot massage, and quiet music. Daily visits will last for the duration of the illness and 7 days following the illness end. Illness end is defined as the last day of illness treatment (e.g., last day of antibiotics) or monitoring (e.g., last day on nursing "24-hour report"). During
Period: Overall Study
Arm/Group | Delirium-prevention Group | Usual Care Group
Started | 114 | 105
Completed | 114 | 105
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Delirium-prevention Group | Usual Care Group | Total
Number analyzed (Participants) | 114 | 105 | 219
Age, Continuous [Mean (Standard Deviation); unit: years] | 82.67 (1.54) | 80.64 (1.34) | 81.69 (1.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 71 | 143
  Male | 42 | 34 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 25 | 65
  Not Hispanic or Latino | 74 | 80 | 154
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 50 | 47 | 97
  White | 59 | 58 | 117
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Cognitive function [Mean (Standard Deviation); unit: units on a scale] — Brief Interview of Mental Status; Score range = 0-15; Higher score = Better mental status function
  units on a scale | 7.95 (.49) | 9.70 (.44) | 8.79 (.44)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Delirium
Description: Confusion Assessment Method (CAM)
Time Frame: During acute condition, up to 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Delirium-prevention Group | Usual Care Group
Number analyzed (Participants) | 114 | 105
Participants | 41 | 33

2. Secondary Outcome: Physical Function at 1 Month
Description: Minimum Data Set Activities of Daily Living scale; Scale range = 0-28; Higher score = Worse activities of daily living function; Outcome measure at 1 month may be adjusted for outcome measure at baseline
Time Frame: Baseline and 1 month
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Delirium-prevention Group | Usual Care Group
Number analyzed (Participants) | 114 | 105
units on a scale | 16.05 (1.13) | 14.27 (1.23)

3. Secondary Outcome: Cognitive Function at 1 Month
Description: Minimum Data Set Cognitive Performance Scale; Scale range = 0-6; Higher scores = Worse cognitive performance; Outcome measure at 1 month may be adjusted for outcome measure at baseline
Time Frame: Baseline and 1 month
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Delirium-prevention Group | Usual Care Group
Number analyzed (Participants) | 114 | 105
units on a scale | 2.06 (.20) | 1.47 (.13)

4. Secondary Outcome: Number of Participants Admitted to Hospital
Time Frame: Up to 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Delirium-prevention Group | Usual Care Group
Number analyzed (Participants) | 114 | 105
Participants | 18 | 19

ADVERSE EVENTS:
Time Frame: 30 days
Description: Fall
Arm/Group | Delirium-prevention Group | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 6/114 | 8/105
Serious Adverse Events (participants affected / at risk) | 18/114 | 19/105
Other Adverse Events (participants affected / at risk) | 30/114 | 16/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delirium-prevention Group (N=114) | Usual Care Group (N=105)
Hospital admission (General disorders) | 18 (22) | 19 (19)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delirium-prevention Group (N=114) | Usual Care Group (N=105)
Fall (General disorders) | 30 (47) | 16 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-11): https://cdn.clinicaltrials.gov/large-docs/79/NCT02994979/Prot_SAP_000.pdf